CLINICAL TRIAL: NCT04983485
Title: Investigation of Respiratory Muscle Activations During Stable Threshold Load and Increasing Threshold Load Endurance Tests in Individuals With COPD
Brief Title: Respiratory Muscle Activations During Stable Threshold Load and Increasing Threshold Load Endurance Tests in COPD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ceyhun Topcuoğlu, Research Assistant, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-CT-02
Record Dates: First submitted 2021-07-09; First posted 2021-07-30 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Surface Electromyography; Ventilation; Respiratory Endurance Test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: Individuals who were diagnosed with COPD by Bolu Abant İzzet Baysal University Medical Faculty Chest Diseases Department and referred to Bolu Abant İzzet Baysal University Health Sciences Faculty Physiotherapy and Rehabilitation Department will be included in the study.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Respiratory muscle electromyographic activations of individuals will be evaluated during the test while breathing rapidly and deeply from the beginning of the constant threshold load endurance test and the increasing threshold load endurance test until the end of the test, and at rest. Respiratory muscle endurance will be evaluated with constant threshold load endurance test and increasing threshold load endurance test, respiratory functions with pulmonary function test, respiratory muscle strength with intraoral pressure measurement device, health condition disorder with Chronic Obstructive Pulmonary Disease Assessment Scale, dyspnea with Modified Medical Research Council Dyspnea Scale and Modified Borg Scale. Participants' names, anthropometric measurements, demographic data, contact information and medical history will be collected and recorded with the patient anamnesis form.

SUMMARY:
In the literature, it has been observed that there is an increase in respiratory muscle activity in individuals with COPD due to the increase in respiratory workload and in response to the loads given by respiratory muscle training devices. However, no study has been found in the literature comparing the activation of respiratory muscles during constant threshold load endurance test and increasing threshold load endurance test performed with respiratory muscle training devices, which are important for respiratory muscle function evaluation. With this planned study, it is aimed to contribute to the literature by examining the changes in muscle activation during the constant threshold load and increasing threshold load endurance tests where different workloads are given and by comparing these changes.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common, preventable and treatable disease characterized by persistent respiratory symptoms and airway limitation due to airway and/or alveolar abnormality that is affected by many factors that cause abnormal lung development resulting from exposure to harmful gases or particles. COPD is known as the fourth most common cause of death in the world and is expected to rise to third place by the end of 2020. Physiopathological changes such as airflow limitation, bronchial fibrosis, increased airway resistance, ciliary dysfunction, gas exchange abnormalities and air trapping occur in COPD. While smoking is the most common risk factor in COPD; Occupational dust and chemicals, air pollution, lung growth and development, genetic predisposition such as age and gender, and exposure to environmental effects. Symptoms such as shortness of breath (dyspnea), cough, and sputum are common in COPD. In addition to pulmonary changes such as an increase in respiratory workload in individuals with COPD, there are also extrapulmonary changes such as respiratory muscle dysfunction.

respiratory muscle dysfunction; It is a decrease in respiratory muscle strength, endurance, or both, resulting from factors such as elongated diaphragm fibers, increased respiratory workload, changes in muscle mass and abdominal weight. Strength is defined as the muscle's capacity to produce power, while endurance is defined as the muscle's ability to sustain a given force over time (the capacity to resist fatigue). Loss of strength and/or endurance contributes to diaphragm weakness and impaired performance. Today, respiratory muscle strength parameters (MIP, MEP) are widely used in the evaluation of respiratory muscle function. However, evaluation of respiratory muscle endurance is more effective than respiratory muscle strength in the evaluation of submaximal respiratory muscle contraction, which is valid for daily activities, and in the clinical, functional and prognostic evaluation of respiratory muscles. Respiratory muscle endurance can be measured with constant threshold load and increased threshold load endurance tests. The imbalance between the function of the respiratory muscles and the respiratory workload they face chronically plays an important role in the formation of dyspnea and hypercapnia. Neural respiratory impulse (NRD), which is indirectly measured by electromyogram (EMG) of respiratory muscles, has attracted attention as a potential physiological marker indicating clinical deterioration due to imbalance between workload and capacity of respiratory muscles. The neural respiratory drive (NRD) is the output of the brainstem respiratory centers. NRD is not affected by the patient's will, is associated with symptoms such as dyspnea, and is usually increased in COPD.

Mechanical abnormalities such as airflow obstruction, static and dynamic hyperinflation, and intrinsic positive end-expiratory pressure increase the load on respiratory muscles in individuals with COPD. Inspiratory muscle contraction is impaired as a result of pressure changes, muscle shortening, increased contraction rate, change in geometry, and decreased compliance of the respiratory system. As a result, an increase in muscle activation and NRD is observed. Those with severe COPD require significantly higher muscle activations, both electrical and mechanical, to breathe and overcome the respiratory workload than those with mild to moderate COPD. In individuals with COPD, NRD increases when the load on the respiratory muscles increases as a result of an increase in respiratory workload, a decrease in capacity, or a combination of both. Studies have shown that, in addition to respiratory workload, workloads given with respiratory muscle training devices lead to an increase in the activation of respiratory muscles.

In the literature, it has been observed that there is an increase in respiratory muscle activity in individuals with COPD due to the increase in respiratory workload and in response to the loads given by respiratory muscle training devices. However, no study has been found in the literature comparing the activation of respiratory muscles during constant threshold load endurance test and increasing threshold load endurance test performed with respiratory muscle training devices, which are important for respiratory muscle function evaluation. With this planned study, it is aimed to contribute to the literature by examining the changes in muscle activation during the constant threshold load and increasing threshold load endurance tests where different workloads are given and by comparing these changes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with chronic obstructive pulmonary disease
* Be between the ages of 40-65
* No medication changes due to acute exacerbation for at least three weeks
* Be stable
* Volunteering to participate in research
* To cooperate
* Patients with written consent form
* Healthy individuals in a similar age range without a diagnosed disease and symptoms will be included

Exclusion Criteria:

* Those with a history of chronic obstructive pulmonary disease exacerbations
* Individuals with orthopedic disease
* Individuals with neurological disease
* Individuals with other co-existing lung and systemic diseases other than chronic obstructive pulmonary disease
* Those who have had major surgery in the past few months
* Individuals with a history of recurrent significant clinical infections
* Have cognitive problems
* Having had unstable angina,
* Previous Myocardial Infarction
* Individuals with severe congestive heart failure refractory to medical therapy, individuals with uncontrolled hypertension
* Individuals with cancer

Ages: 40 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chronic obstructive pulmonary disease (COPD) is a common, preventable and treatable disease characterized by persistent respiratory symptoms and airway limitation due to airway and/or alveolar abnormality resulting from exposure to harmful gases or particles and many factors that cause abnormal lung development.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2023-06-25 (Estimated); Primary Completion 2023-07-25 (Estimated); Study Completion 2023-08-25 (Estimated)

PRIMARY OUTCOMES:
Surface Electromyography | 45 minutes
  Activation of respiratory muscles will be performed with a surface Electromyography (EMG) device. The measurement will be performed by placing Electromyography (EMG) electrodes on the motor points of the respiratory muscles. Increased respiratory muscle activations indicate that respiratory muscles are used more; The decrease in respiratory muscle activations indicates that the respiratory muscles are used less.

SECONDARY OUTCOMES:
Incremental Threshold Load Endurance Test | 10 minutes
  Respiratory muscle endurance will be measured with an incremental threshold load respiratory muscle endurance test. The respiratory muscle endurance test will be performed using a respiratory muscle training device. Endurance test is performed by breathing rapidly and deeply against the respiratory muscle training device of the individual. The individual should continue the test as long as possible. A high respiratory muscle endurance score indicates good respiratory muscle function; A low score indicates respiratory muscle dysfunction.
Sustained Threshold Load Endurance Test | 10 minutes
  Respiratory muscle endurance will be measured with an sustained threshold load respiratory muscle endurance test. The respiratory muscle endurance test will be performed using a respiratory muscle training device. Endurance test is performed by breathing rapidly and deeply against the respiratory muscle training device of the individual. The individual should continue the test as long as possible. A high respiratory muscle endurance score indicates good respiratory muscle function; A low score indicates respiratory muscle dysfunction.
Pulmonary Function Test: | 5 minutes
  Pulmonary function test will be performed with a spirometer according to the criteria of the American Thoracic Society and the European Respiratory Society. While the decrease in pulmonary function test parameters shows worsening of lung functions; parameters in the normal range indicate good lung functions.
Measurement of Maximal Inspiratory Pressure | 5 minutes
  Maximal Inspiratory Pressure will be measured with an intraoral pressure measuring device. Maximal Inspiratory Pressure reflects respiratory muscle strength. An increase in Maximal Inspiratory Pressure indicates high respiratory muscle strength; A low Maximal Inspiratory Pressure value indicates respiratory muscle weakness.
Chronic Obstructive Pulmonary Disease Assessment Test | 2 minutes
  Chronic Obstructive Pulmonary Disease Assessment Test is an eight-item scale measuring health status in Chronic Obstructive Pulmonary Disease. This scale is used to determine the health status of individuals with Chronic Obstructive Pulmonary Disease all over the world. Each question is scored between 0-5 and a total score between 0 and 40 is given. A score of 0 represents the best and a score of 40 represents the worst state of health.
Modified Medical Research Council Dyspnea Scale | 2 minutes
  It is a 5-item scale scored between 0-4 for individuals' shortness of breath. Evaluates dyspnea and activity limitation in individuals with COPD
Modified Borg Scale (MBS) Çeviri sonuçları Modified Borg Scale (MBS): | 2 minutes
  It is a 5-item scale scored between 0-4 for individuals' shortness of breath. Evaluates dyspnea and activity limitation in individuals with chronic obstructive pulmonary disease. An increase in the score indicates an increase in shortness of breath.

IPD SHARING:
Plan to Share IPD: No